CLINICAL TRIAL: NCT02414685
Title: A Treatment Strategy of the Use of 1st Line Chemotherapy in Patients With Poor-Prognosis Disseminated Non-Seminomatous Germ Cell Tumors Based on Tumor Marker Decline: A Phase II Trial of Paclitaxel, Ifosfamid and Cisplatin Regimen.
Brief Title: First Line TIP in Poor Prognosis TGCTs.
Acronym: TIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Slovakia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCTSK003
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Germ Cell Tumor
Keywords: poor-prognosis germ cell cancer, paclitaxel, ifosfamid and cisplatin regimen, tumor marker decline
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Paclitaxel; Ifosfamide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intravenous chemotherapy (Experimental): TIP regimen:
  * Paclitaxel 250 mg/ m2 iv on day 1
  * Ifosfamide 1,2 g/ m2/ day iv x 5 days
  * Cisplatin 20 mg/ m2/ day iv x 5 days
  Interventions: Drug: Paclitaxel; Drug: Ifosfamide; Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel — paclitaxel, ifosfamide, cisplatin until progression, unacceptable toxicity, complete response or inability of the subject to comply with study requirements
  Other Names: paclitaxel ebewe
Drug: Ifosfamide — paclitaxel, ifosfamide, cisplatin until progression, unacceptable toxicity, complete response or inability of the subject to comply with study requirements
  Other Names: ifosfamide-holoxan
Drug: Cisplatin — paclitaxel, ifosfamide, cisplatin until progression, unacceptable toxicity, complete response or inability of the subject to comply with study requirements
  Other Names: cisplatin-hospira

SUMMARY:
TIP in the 1st line treatment of GCTs patients with unfavorable decline of serum tumor markers after 1 cycle of the BEP regimen.TIP will be administered to the patient until progression, unacceptable toxicity, complete response or inability of the subject to comply with study requirements.

DETAILED DESCRIPTION:
Cycle 1: BEP regimen

Serum tumor markers at day 18-21:

•Patients with an unfavorable pattern of tumor marker decrease after 1 cycle of BEP will receive 4 more cycles of TIP.

TIP regimen:

* Taxol 250 mg/ m2 iv on day 1
* Ifosfamid 1,2 g/ m2/ day iv x 5 days
* Cisplatin 20 mg/ m2/ day iv x 5 days One cycle of therapy consists of 22 days. Estimated duration of treatment: Until progression, unacceptable toxicity, complete response or inability of the subject to comply with study requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 16 years.
* Evidence of NSGCT based on histologic examination or based on clinical evidence and high serum HCG or AFP levels (in case of clinical emergency, therapy can be started before pathologic sample is obtained if tumor markers are very elevated)
* Testicular, retroperitoneal, or mediastinal primary site.
* Evidence of disseminated disease (clinical stages II or III).
* Disease classified as poor prognosis according to IGCCCG criteria:
* Primary mediastinal NSGCT or
* Non-pulmonary visceral metastases or
* HCG > 50,000 UI/l, or AFP > 10,000 ng/ml, or LDH > 10 times the upper normal value.
* No prior chemotherapy.
* No previous carcinoma, except basal-cell carcinoma of the skin.
* Adequate renal function: measured or calculated creatinine clearance> 60 ml/min.
* Absolute granulocyte count >= 1,500/mm3, platelets >= 100,000 mm3, bilirubine <= 1.5 fold the upper normal value.
* Unfavorable tumor marker decline after 1.cycle of BEP
* Signed informed consent.

Exclusion Criteria:

* Patients infected by the Human Immunodeficiency Virus (HIV).
* Patients who do not fit inclusion criteria.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-04; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Complete response rate | 36 month
  according RECIST criteria version 1.1

SECONDARY OUTCOMES:
Response rate | 36 month
  response rate after chemotherapy
Progression-free survival | 36 month
  expressed as median and as 12-weeks post-treatment initiation continuous progression-free survival rate
Number of adverse events grade III and IV | 36 month
overall survival | 36 months
  Survival will be estimated from the registration date to the date of last follow-up or death. Patients will be followed at least 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mego, Ass.prof, Study Chair — National Cancer Institute, Slovakia
Locations (1):
- National Cancer Institute, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided